CLINICAL TRIAL: NCT03261089
Title: Addressing an Inherent Bias in Neuroprognostication: A Collaboration to Reduce the Impact of Self-fulfilling Prophecy in Cardiac ARrEst
Brief Title: Neuroprognostication Bias: A Collaboration to Reduce the Impact of Self-fulfilling Prophecy in Cardiac ARrEst
Acronym: SPARE
Status: Recruiting | Type: Observational
Sponsor: Boston Medical Center (Other)
Collaborators: University of Florida (Other); Hospital Israelita Albert Einstein (Other); Faculty of Medicine of Ribeirão Preto (FMRP-USP) (Other); University of Sao Paulo General Hospital (Other); Yale University (Other); University of Pennsylvania (Other); University of California, San Francisco (Other); D'Or Institute for Research and Education (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: H-36257, H-45526; R01NS128342 (NIH)
Record Dates: First submitted 2017-08-21; First posted 2017-08-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; neuroprognostication; coma
MeSH Terms: conditions — Heart Arrest; Coma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Unresponsive patients post-cardiac arrest: As early as possible post-resuscitation, patients should undergo a detailed neurologic examination, comprised of a thorough assessment for consciousness and detailed cranial nerve function and motor response assessments. Neurologic assessment scores such as the Full Outline of Unresponsiveness, Glasgow Coma Scale (GCS), and Pittsburgh Cardiac Arrest Category (PCAC) Score will be also be used. On the first assessment (day of cardiac arrest), the PCAC score should be assigned only on the basis of the best neurologic exam in the first 6 hours after ROSC. Patients that are sedated or intubated will have the verbal score of GCS be estimated by a derivation of motor and eye scores. The presence of potential confounders, including core body temperature, medications, and/or intoxicants, as well as metabolic derangements will be noted.

SUMMARY:
Cardiovascular disease remains the leading cause of death in the United States. Mortality rates of cardiac arrest range from 60-85%, and approximately 80% of survivors are initially comatose. Of those who survive, 50% are left with a permanent neurological disability, and only 10% are able to resume their former lifestyle. Early prognosis of comatose patients after cardiac arrest is critical for management of these patients, yet predicting outcome for these patients remains quite challenging.

The primary study objective of SPARE is to assess the value of using a systematic, multi-modal approach for neuroprognostication in the unconscious post-cardiac arrest population. We hypothesize that prognostication using this approach will be significantly improved compared to historical controls. This approach will be novel because:

All patients who are unconscious at least 24 hours post-cardiac arrest, whereas previous studies on neurologic outcome tended to have restrictive inclusion criteria, such as no pre-existing neurologic impairment (e.g. dementia or prior cerebrovascular injury), or included an unduly restrictive population, such as patients with a strictly comatose state.

The prognostic modalities used to assess patients will be applied at specific time points that will maximize their utility.

Patients' families and clinicians will be encouraged to provide adequate time to allow for a delayed recovery, especially in cases of uncertain outcome, thus minimizing the self-fulfilling prophesy bias of early withdrawal of life-sustaining therapies (WLST). This will be particularly pertinent in the comparison of US and Brazil/Italy patients, as the Brazilian and Italian populations are not commonly exposed to premature WLST (as can be the case in the US), one of the major sources of biases in prognostication studies of cardiac arrest due to the self-fulfilling prophecy.

DETAILED DESCRIPTION:
SPARE is a multi-center, international, prospective registry designed to evaluate the use of a multi-modality approach to neuroprognostication after cardiac arrest. Subjects will be evaluated with standard, accepted, and widely available assessment modalities, including clinical examination, neurophysiologic (electroencephalography and evoked potentials (per site standard of care), serum biomarkers (per site standard of care), and neuroimaging testing.

The purpose of this study is to collect data from a prospective large-scale cohort involving cardiac arrest survivors, and the clinical characteristics and prognostic features that affect their neurologic outcome. The ultimate goal is to derive a prediction model for neuroprognostication in cardiac arrest, using multiple clinical modalities that are already clinically in use, but in a standardized fashion. We hypothesize that by using a multimodal approach combining clinical assessment tools obtained at standardized time points, we will improve the accuracy of neuroprognostication in initially unconscious cardiac arrest survivors. The US and non-US populations will be compared, as the non-US population is less exposed to early WLST, thus eliminating the self-fulfilling prophecy bias that has plagued all CA studies to date.

Outcomes will be assessed at discharge, at 3 months post-arrest, 6 months, and annually up to 5 years afterwards. The primary outcome will be the proportion of subjects with good versus poor outcome, with a dichotomized approach of the modified Rankin Scale (mRS): good outcome defined as mRS scores of 0-3, and poor outcome as mRS scores of 4-6. Secondary outcome measures include overall scores on the Cerebral Performance Category Scale (CPC), Cerebral Performance Category - Extended (CPC-E), and Montreal Cognitive Assessment (MOCA) (or Telephone Montreal Cognitive Assessment (T-MOCA)).

ELIGIBILITY:
Inclusion Criteria:

* Initially unconscious following cardiac arrest from any non-perfusing rhythm (i.e., ventricular tachycardia, ventricular fibrillation, pulseless electrical activity, asystole)
* Sustained return of spontaneous circulation (ROSC) as defined by maintained spontaneous circulation for at least 20 minutes after cardiopulmonary resuscitation.

Exclusion Criteria:

- Isolated respiratory arrest without concomitant or ensuing cardiac arrest

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unresponsive patients post-cardiac arrest
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-08-02 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Score (mRS) | 14 days, 3 months post-arrest, 6 months, and annually up to 5 years afterwards
  A 7-point scale that measures the level of disability or impairment. mRS 0-3 is considered a good outcome while mRS is considered a poor outcome

SECONDARY OUTCOMES:
Cerebral Performance Category Scale (CPC) | 14 days, 3 months post-arrest, 6 months, and annually up to 5 years afterwards
  A scale from 1-5 assessing brain function and used to gauge neurological recovery. CPC 1 or 2 is considered good outcome while CPC 3-5 is considered poor outcome
Cerebral Performance Category- Extended (CPC-E) | 14 days, 3 months post-arrest, 6 months, and annually up to 5 years afterwards
  An advanced multi-domain tool used to assess the detailed neurological and functional recovery.
Montreal Cognitive Assessment (MOCA) | 14 days, 3 months post-arrest, 6 months, and annually up to 5 years afterwards
  A Screening tool for cognitive impairment. Score from 0-30
Short Form 36 | 14 days, 3 months post-arrest, 6 months, and annually up to 5 years afterwards
  A 36 item patient reported survey used to measure health status and quality of life.
Glasgow Outcome Scale-Extended (GOS-E) | 14 days, 3 months post-arrest, 6 months, and annually up to 5 years afterwards
  An 8-point scale used to measure global disability and functional outcome

CONTACTS AND LOCATIONS:
Overall Officials: David M Greer, MD MA, Principal Investigator — Boston Medical Center, Neurology; Gisele Sampaio-Silva, MD, Principal Investigator — Hospital Israelita Albert Einstein, Neurology
Locations (8):
- United States (5):
  - University of California, San Francisco, San Francisco, California
  - Yale University, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Boston Medical Center, Boston, Massachusetts
  - University of Pennsylvania, Philadelphia, Pennsylvania
- Brazil (3):
  - Instituto D'Or de Pesquisa e Ensino, Rio de Janeiro
  - Albert Einstein Israelite Hospital, São Paulo
  - Hospital das Clinicas Faculdade de Medicina Ribeirao Preto, São Paulo

IPD SHARING:
Plan to Share IPD: No